CLINICAL TRIAL: NCT05683002
Title: Aronia, Cognition, and Eye Health
Brief Title: Aronia, Cognition, and Eye Health (ACE)
Acronym: ACE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: BioActor B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: BB-04
Record Dates: First submitted 2022-12-08; First posted 2023-01-12 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Cognitive Function
Keywords: Supplementation; Cognition; Cognitive Function

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Block Randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aronia (Experimental): Aronia Melanocarpa supplementation
  Interventions: Dietary Supplement: Aronia supplementation
- Control (Placebo Comparator): Cellulose supplementation
  Interventions: Dietary Supplement: Cellulose supplementation

INTERVENTIONS:
Dietary Supplement: Aronia supplementation — As described in experimental arm
  Arms: Aronia
Dietary Supplement: Cellulose supplementation — As described in placebo comparator arm
  Arms: Control

SUMMARY:
There is great interest in improving cognitive performance and eye health as working from home becomes more prominent. Working from home as well as stress in the workplace is an increasing problem. Students and work professional can therefore benefit from improved attention and thus performance in academic and other work environments. A completely natural supplement with aronia melanocarpa extract could be a promising way to naturally improve cognitive performance

DETAILED DESCRIPTION:
The shift of on-site education/working to online education/working has had a detrimental impact on motivation to study or work and ultimately on mental health. Moreover, online education has been shown to have a negative effect on concentration, learning, and academic performance. Stress in the workplace is an increasing problem, leading to decreased productivity and overall well-being of working adults. Consequently, there is a great interest in improving cognitive performance, including memory and attention.

Previous studies in young adults have mainly focused on acute or short-term (e.g. 1 week) effects of anthocyanin supplementation on cognitive performance. The research hypothesis of the current study is that long term (6 weeks) AME supplementation affects domains of cognitive performance in a randomized, double-blind, placebo controlled, cross-over study in healthy young adults (18-35 years old).

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women, aged between 18-35 years
* BMI between 18-30 kg/m2
* Systolic blood pressure < 160 mmHg and diastolic blood pressure < 100 mmHg
* Stable body weight (weight gain or loss < 3 kg in the past three months)
* Willingness to give up being a blood donor from 8 weeks before the start of the study, during the study and for 4 weeks after completion of the study
* No difficult venipuncture as evidenced during the screening visit

Exclusion Criteria:

* Smoking or smoking cessation < 12 months
* Contact lens wearers
* Past refractive surgery
* Severe medical conditions, including asthma, chronic obstructive pulmonary disease (COPD), kidney failure, auto-inflammatory diseases, rheumatoid arthritis, diabetes mellitus, cardiovascular disease
* Use of dietary supplements or medication affecting the main outcomes of the study
* Use of an investigational product within another biomedical intervention trial within the previous month
* Familial hypercholesterolemia
* Abuse of drugs
* More than 3 alcoholic consumptions per day

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-12-08 (Actual); Primary Completion 2024-07-26 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Cognitive Function | After 6 weeks of supplementation
  Quantified through the Cambridge Neuropsychological Test Automated Battery (CANTAB). Focus on attention/psychomotor speed, memory, and executive function

SECONDARY OUTCOMES:
Eye Health | At baseline and after 6 weeks of supplementation
  Tear fluid collection (volume)
Subjective Eye Fatigue | At baseline and after 6 weeks of supplementation
  Subjective Eye Fatigue Questionnaire
Vascular Function | At baseline and after 6 weeks of supplementation
  Fundus photography

CONTACTS AND LOCATIONS:
Overall Officials: Jogchum Plat, Prof, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No